CLINICAL TRIAL: NCT06159049
Title: Clinical Translation of a Novel FAPI Dimer [68Ga]Ga-LNC1013
Status: Completed | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: PETcenter
Record Dates: First submitted 2023-09-17; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-09

CONDITIONS: Gastrointestinal Cancer
Keywords: FAPI dimer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI dimer(68Ga-LNC1013) — 68Ga-LNC1013 was evaluated in a pilot clinical PET imaging study involving seven patients with gastrointestinal cancer.

SUMMARY:
Fibroblast activation protein (FAP) emerges as a highly promising target for cancer diagnostic imaging and targeted radionuclide therapy. To exploit the therapeutic potential of current FAP inhibitors (FAPIs), this study presented the design and synthesis of a series of FAPI dimers to increase tumor uptake and retention. Preclinical evaluation and a pilot clinical PET imaging study were conducted to screen the lead compound with the potential for radionuclide therapy.

DETAILED DESCRIPTION:
Three new FAPI dimers were synthesized by linking two quinoline-based FAPIs with different spacers. The in vitro binding affinity and preclinical small animal PET imaging of the compounds were compared with their monomeric counterparts, FAPI-04 and FAPI-46. The lead compound, 68Ga-LNC1013, was then evaluated in a pilot clinical PET imaging study involving seven patients with gastrointestinal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or clinically confirmed and/or suspicious of gastrointestinal cancer.
2. Signed informed consent.

Exclusion Criteria:

1. pregnancy;
2. breastfeeding;
3. any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Claustrophobia (unable to accept PET/CT scanning)
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Number of discrepancies between [68Ga]Ga-LNC1013 and 68Ga-FAPI-46 or 18F-FDG PET scans | 5 months
  Compare the diagnostic performance between [68Ga]Ga-LNC1013 and 68Ga-FAPI-46 or 18F-FDG in patients with gastrointestinal cancer
SUVmaxFAPI and SUVmaxFDG for each target (Standardized Uptake Value) | 5 months
  Comparison of 68Ga]Ga-LNC1013, 68Ga-FAPI-46 and 18F-FDG Standardized Uptake Value in the primary tumor and possible metastases

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Hu, Dr, Study Chair — Xiangya Hospital, Central South University, Changsha, P.R. China
Locations (1):
- Jian Li, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No